CLINICAL TRIAL: NCT06353893
Title: Postoperative MRI Evaluation of the Integrity Bio-inductive Implant Augmentation of Rotator Cuff Tears of the Shoulder
Brief Title: MRI Evaluation of Integrity Implant for Rotator Cuff Tears
Status: Active, not recruiting | Type: Observational
Sponsor: Foundation for Orthopaedic Research and Education (Other)
Collaborators: Anika Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Integrity-001
Record Dates: First submitted 2024-03-13; First posted 2024-04-09 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Anika Integrity Implant System — The implant is a porous, flexible construct knitted using HYAFF® fibers and designed to support cell infiltration and regenerative healing. HYAFF is Anika's proven and proprietary esterified HA technology that resorbs over time as tissue remodels. Integrity is inherently strong and can be confidently manipulated arthroscopically, which offers a truly unique and differentiated solution for shoulder surgeons to treat rotator cuff tears.

SUMMARY:
The goal of this observational study is to evaluate the effectiveness and safety of the Integrity bio-inductive implant in treating partial and full thickness rotator cuff tears. The main questions it aims to answer are:

* How does the application of the Integrity implant affect patient-reported outcome measures (PROMs) such as ASES, SANE, and PROMIS?
* What are the imaging characteristics of the rotator cuff tears at 3 and 6 months postoperatively when using the Integrity implant?

Postoperative MRIs will be obtained from 10 consecutive patients who have undergone rotator cuff repair using the Integrity implant at 3 and 6 months after surgery. Participants include those with partial and full thickness tears treated with different surgical techniques involving the implant. They may receive either isolated onlay use of the graft for partial tears or augmentation of a standard single or double row repair with the graft applied to the superior surface of the repair.

DETAILED DESCRIPTION:
The aim of this prospective, non-randomized, open-label, single-arm study is to evaluate the safety and effectiveness of the newly FDA-cleared Integrity graft for various types of rotator cuff repairs. This study incorporates preoperative assessments as well as follow-up assessments at 3 months and 6 months postoperatively. The primary objective is to document the safety profile of the Integrity graft by monitoring device-related adverse events throughout the study duration. Additionally, the study aims to assess the post-market effectiveness of the Integrity implant using patient-reported outcome measures and establish normal or standard findings on MRI to aid surgeons in clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Rotator cuff tear (both partial and full thickness) treated with Integrity bio-inductive implant augmentation to the superior surface of partial rotator cuff tears or the superior aspect of rotator cuff repairs (both single or double row);
* Subject can read and understand the ICF and has voluntarily provided written informed consent.

Exclusion Criteria:

* Conditions which, in the opinion of the Principal Investigator, may limit the subject's ability or willingness to follow post- operative care or study instructions;
* If patient is pregnant;
* Subject conditions which may hinder the healing process;
* Subject is a prisoner or member of another vulnerable population.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be recruited from patients with a history of rotator cuff repair surgery one to 83 days (about 2 and a half months) before the screening.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
MRI Assessment of Adverse Events and Structural Integrity | 3 and 6 months after index procedure
  The primary endpoint of this study is the adverse events rate and structural failure rate of the rotator cuff repair, determined by MRI, at 3 months and 6 months following use of the Anika Integrity implant system.

SECONDARY OUTCOMES:
Effectiveness Evaluation with PROMIS outcome tool | 3 months after index procedure
  The secondary endpoints of the study include evaluating PROMIS scores (assessing various aspects of quality of life in a questionnaire which is scored)
Effectiveness Evaluation with PROMIS tool | 6 months after index procedure
  The secondary endpoints of the study include evaluating PROMIS scores (assessing various aspects of quality of life)
Effectiveness Evaluation with SANE score | 3 months after index procedure
  The secondary endpoints of the study include evaluating SANE scores: Single assessment numeric rating scale of 0-10 with 0 being NO pain and 10 being worst or severe pain (patients' perceived improvement)
Effectiveness Evaluation with SANE score | 6 months after index procedure
  The secondary endpoints of the study include evaluating SANE scores: Single assessment numeric rating scale of 0-10 with 0 being NO pain and 10 being worst or severe pain (patients' perceived improvement)
Effectiveness Evaluation with ASES rating scale | 3 months after index procedure
  The secondary endpoints of the study include evaluating ASES rating scale (for shoulder function and pain) ASES is a mixed-outcome reporting tool, meaning it consists of a physician-rated and patient-rated questionnaire. The patient-rated questionnaire focuses on joint pain, instability and activities of daily living.
Effectiveness Evaluation with ASES rating scale | 6 months after index procedure
  The secondary endpoints of the study include evaluating ASES rating scale (for shoulder function and pain)ASES is a mixed-outcome reporting tool, meaning it consists of a physician-rated and patient-rated questionnaire. The patient-rated questionnaire focuses on joint pain, instability and activities of daily living.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation for Orthopaedic Research and Education, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No